CLINICAL TRIAL: NCT02640560
Title: One-year Survey of Anaphylaxis in Outpatient Children Allergic to Peanuts, Walnuts/Hazelnuts, Shellfish
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 10/2012
Record Dates: First submitted 2015-12-09; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Food Allergy
Keywords: Children; Allergy; Peanuts; Hazelnuts; Walnuts; Mollusks; Shellfish; Food
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with food allergy: Children with food allergy to nuts, hazelnuts, walnuts, shellfish and mollusks (1-14 years old).
  The Parents of the cases children will compile a Food allergy questionnaire
  Interventions: Other: Food allergy questionnaire
- Healthy Children: Healthy Children (1-14 years old) The Parents of the control children will compile a Control questionnaire
  Interventions: Other: Control Questionnaire

INTERVENTIONS:
Other: Food allergy questionnaire — The Parents of the cases children will compile a questionnaire including questions about general information on the family, on life and food habits, on indoor environment, on health status, on clinical aspects of the allergy, on the access to diagnostic and treatment resources
  Groups: Children with food allergy
Other: Control Questionnaire — The Parents of the control children will compile a questionnaire including questions about general information on the family, on life and food habits and on indoor environment.
  Groups: Healthy Children

SUMMARY:
In Italy, few data about anaphylaxis due to peanuts in pediatric age are available, conversely data about walnuts/hazelnuts, shellfish/mollusks anaphylaxis have not yet been collected.

Children with physician-confirmed food allergy to peanuts, walnuts/hazelnuts and shellfish/mollusks will be recruited from 9 allergy clinics located in the Italian Territory (Bologna, Lecce, Napoli, Palermo, Parma, Pavia, Roma, Torino, Trento).

Parent of food allergic children will compile a food allergy questionnaire (questions about general information on the family, on life and food habits, on indoor environment, on health status, on clinical aspects of the allergy, on the access to diagnostic and treatment resources).

Parent of healthy children will compile a control questionnaire (questions about general information on the family, on life and food habits and on indoor environment) The 1-year survey will determine the frequency of anaphylaxis in allergic outpatient children.

ELIGIBILITY:
Inclusion criteria

* Cases: 0-14 years old patients with food allergy to peanuts, walnuts/hazelnuts, shellfish/mollusks.
* Controls: 0-14 years old subjects without allergy to peanuts, walnuts/hazelnuts, shellfish/mollusks.

Exclusion criteria

* Patients/subjects in acute phase of disease or with not controlled chronic pathologies;
* missing written informed consent by parents

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 200 Italian children with or without food allergy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Anaphylaxis in 1 year | 1 year
  To determine the frequency of anaphylaxis in allergic outpatient children